CLINICAL TRIAL: NCT00944710
Title: Augmenting Atropine Treatment for Amblyopia in Children 3 to < 8 Years Old
Acronym: ATS16
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-144; 2U10EY011751 (NIH)
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Amblyopia
Keywords: Amblyopia; atropine; Plano lens
MeSH Terms: conditions — Amblyopia | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intensified treatment (Active Comparator): Weekend atropine 1% with plano lens over the sound eye
  Interventions: Drug: Atropine; Device: Plano lens
- Control (Active Comparator): Weekend atropine 1%
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — Weekend atropine 1%
  Arms: Intensified treatment
Device: Plano lens — plano lens over the sound eye
  Arms: Intensified treatment
Drug: Atropine — Weekend atropine 1%
  Arms: Control

SUMMARY:
This study is designed to evaluate the effectiveness of adding a plano lens to weekend atropine after visual acuity has stabilized with weekend atropine but amblyopia is still present. Children ages 3 to <8 years with visual acuity of 20/50 to 20/400 in the amblyopic eye will be enrolled in a run-in phase with weekend atropine until no improvement, followed by randomization of eligible patients to weekend atropine treatment with a plano lens over the sound eye versus without a plano lens over the sound eye. The primary objective is to determine if adding a plano lens to weekend atropine will improve visual acuity in patients with amblyopia still present after visual acuity has stabilized with initial treatment.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Both patching and atropine are accepted treatment modalities for the management of moderate amblyopia in children.1 Many practitioners prescribe weekend atropine as initial therapy for amblyopia. However, many children fail to achieve normal visual acuity in the amblyopic eye after treatment with this regimen. In a randomized trial conducted by PEDIG comparing atropine regimens, 58 of 83 patients with moderate amblyopia (70%) had amblyopic eye visual acuity of 20/32 or worse after 4 months of treatment with weekend atropine.2 In another PEDIG randomized trial comparing atropine with a plano lens versus without a plano lens for initial treatment of amblyopia, 60 of 84 patients with moderate amblyopia (71%) had amblyopic eye visual acuity of 20/32 or worse after 16 weeks of treatment with weekend atropine.3 When improvement stops after initial therapy and amblyopia is still present, treatment options include increasing the dosage of current treatment, switching to another treatment, maintaining the same treatment and dosage, or combining treatments. Many clinicians will add a plano lens over the sound eye to atropine treatment, in part because families using atropine have become comfortable with its use. This option is limited to children with hypermetropia in the sound eye. However, it is unknown whether adding a plano lens over the sound eye will improve amblyopic eye visual acuity more than continuing atropine alone in patients who have shown no improvement after initial treatment with atropine. In a PEDIG randomized trial comparing patching to atropine for initial treatment of amblyopia, a plano lens was prescribed for the sound eye for 55 patients who had not improved to 20/30 or at least 3 lines after 4 months of daily atropine use.1, 4 Their mean acuity improvement prior to using the plano lens was 1.0 line, compared with 1.6 lines after prescribing the plano lens. We are unaware of any reports of the response of treatment of amblyopia still present after initial treatment with weekend atropine.

ELIGIBILITY:
Inclusion Criteria:

Major Eligibility Criteria for Run-in Phase

* Age 3 to < 8 years
* Amblyopia associated with strabismus, anisometropia, or both
* Visual acuity in the amblyopic eye between 20/50 and 20/400 inclusive
* Visual acuity in the sound eye 20/32 or better and inter-eye acuity difference >3 logMAR lines
* Amblyopia treatment within the past 6 months subject to the following stipulations:

  * No more than 6 weeks of any amblyopia treatment other than spectacles (except for patients being treated with atropine who are entering the study on treatment)
  * No simultaneous treatment with patching and atropine
  * No use of atropine in combination with the sound eye spectacle lens reduced by more than 1.50 D
  * Maximum level of treatment within the past 6 months:

    * Patching: up to 2 hours daily
    * Atropine: up to once daily
* Wearing spectacles with optimal correction (if amblyopic eye acuity is 20/80 or better, then VA must be stable in glasses; if amblyopic eye acuity is 20/100 or worse, then spectacles and atropine can be initiated simultaneously).
* Hypermetropia and spectacle correction in sound eye of +1.50 D or more

Eligibility Criteria for Randomization:

* Amblyopic eye acuity of 20/40 to 20/160 with an inter-ocular difference of >2 lines, or amblyopic eye acuity of 20/32 with 3 lines of IOD.
* Compliance with weekend atropine treatment based on investigator judgment.

Exclusion Criteria:

* Currently using vision therapy or orthoptics
* Ocular cause for reduced visual acuity (nystagmus per se does not exclude the patient if the above visual acuity criteria are met)
* Prior intraocular or refractive surgery
* Known allergy to atropine or other cycloplegic drugs
* Down Syndrome present

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2009-08; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David K. Wallace, M.D., Study Chair — Duke University Eye Center
Locations (2):
- United States (2):
  - Southern California College of Optometry, Fullerton, California
  - Duke University Eye Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website at http://pedig.jaeb.org/Studies.aspx?RecID=30

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group; Wallace DK, Lazar EL, Repka MX, Holmes JM, Kraker RT, Hoover DL, Weise KK, Waters AL, Rice ML, Peters RJ. A randomized trial of adding a plano lens to atropine for amblyopia. J AAPOS. 2015 Feb;19(1):42-8. doi: 10.1016/j.jaapos.2014.10.022. PMID 25727586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2009 and August 2013, 73 participants from 20 sites were randomly assigned to either augmenting weekend atropine by changing the lens over the fellow eye to plano (n=33) or continuing with weekend atropine with best spectacle correction (n=40).
Pre-assignment Details: Prior to being considered for the randomized trial, participants who had not completed at least 12 weeks of atropine were enrolled into a run-in phase and treated with weekend atropine 1% ophthalmic solution and spectacles based upon a recent cycloplegic refraction, with follow up every 6 weeks until no improvement
Period: 10-week Primary Outcome
Arm/Group | Control | Intensified Treatment
Started | 40 | 33
Completed | 40 | 33
Not Completed | 0 | 0
Period: 12-week Visit (Off-treatment)
Arm/Group | Control | Intensified Treatment
Started | 40 | 33
Completed | 40 | 33
Not Completed | 0 | 0
Period: Additional Post 10-week Primary Outcome
Arm/Group | Control | Intensified Treatment
Started | 40 | 33
Eligible to Enter Post 10-week Phase | 24 | 26
Completed | 23 | 22
Not Completed | 17 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intensified Treatment | Total
Number analyzed (Participants) | 40 | 33 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 40 | 33 | 73
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (1.5) | 5.8 (1.4) | 5.8 (1.4)
Age, Customized [Number; unit: participants] — Baseline age reflects age at randomization.
  The age eligibility requirement at enrollment was 3 to <8 years old; however, four participants (2 in each group) were <8 years old at time of enrollment into the run-in phase and ≥ 8 years old at time of randomization (8.0 and 8.1 in the atropine only group, and 8.1 and 8.3 in the atropine plus plano lens group).
  participants
    3 to <4 years | 5 | 4 | 9
    4 to <5 years | 8 | 6 | 14
    5 to <6 years | 9 | 9 | 18
    6 to <7 years | 7 | 5 | 12
    >=7 years | 11 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 18 | 14 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  White | 33 | 29 | 62
  African American | 3 | 1 | 4
  Hispanic | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 40 | 33 | 73
Duration of Atropine Treatment Prior to Randomization [Number; unit: participants]
  12 to <15 weeks | 11 | 5 | 16
  15 to <21 weeks | 6 | 9 | 15
  21 to <27 weeks | 13 | 9 | 22
  27 to 84 weeks | 10 | 10 | 20
Duration of Atropine Treatment Prior to Randomization [Mean (Standard Deviation); unit: weeks] | 24.0 (11.2) | 26.4 (14.6) | 25.0 (12.8)
Cause of Amblyopia [Number; unit: participants] — Amblyopia associated with strabismus (comitant or incomitant), anisometropia, or both:
  Criteria for strabismus: At least one of the following:
  1. Heterotropia at distance and/or near fixation on examination (with or without spectacles)
  2. History of strabismus surgery
  3. Documented history which is no longer present (which in the judgement of the investigator could have caused amblyopia)
  Criteria for anisometropia: At least one of the following:
  1. At least 0.50 D difference between eyes in spherical equivalent
  2. At least 1.50 D different between eyes in astigmatism in any meridian
  participants
    Strabismus | 9 | 13 | 22
    Anisometropia | 10 | 6 | 16
    Strabismus and Anisometropia | 21 | 14 | 35
Distance Visual Acuity in the Amblyopic Eye at Randomization [Number; unit: participants] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  participants
    20/160 | 2 | 1 | 3
    20/125 | 2 | 2 | 4
    20/100 | 5 | 1 | 6
    20/80 | 2 | 6 | 8
    20/63 | 9 | 8 | 17
    20/50 | 7 | 8 | 15
    20/40 | 11 | 6 | 17
    20/32 | 2 | 1 | 3
Distance Visual Acuity in the Amblyopic Eye at Randomization [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  logMAR | 0.48 (0.19) | 0.48 (0.16) | 0.48 (0.18)
Distance Visual Acuity in the Fellow Eye at Randomization [Number; unit: participants] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  participants
    20/32 | 5 | 6 | 11
    20/25 | 13 | 9 | 22
    20/20 | 16 | 13 | 29
    20/16 | 6 | 5 | 11
Distance Visual Acuity in the Fellow Eye at Randomization [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured without cycloplegia using the participant's optimal spectacle correction by a study-certified tester using the ATS-HOTV protocol on the Electronic Visual Acuity Tester.
  logMAR | 0.04 (0.09) | 0.05 (0.10) | 0.05 (0.09)
Interocular Eye Visual Acuity Difference at Randomization [Mean (Standard Deviation); unit: logMAR lines] | 4.4 (1.8) | 4.4 (1.7) | 4.4 (1.7)
Spherical Equivalent Refractive Error in Amblyopic Eye at Enrollment [Number; unit: participants]
  0 to <+1.00 D | 0 | 0 | 0
  +1.00 to <+2.00 D | 0 | 1 | 1
  +2.00 to <+3.00 D | 1 | 1 | 2
  +3.00 to <+4.00 D | 6 | 5 | 11
  +4.00 D or more | 33 | 26 | 59
Spherical Equivalent Refractive Error in Amblyopic Eye at Enrollment [Mean (Standard Deviation); unit: diopters] | 5.73 (1.62) | 5.84 (1.89) | 5.78 (1.74)
Spherical Equivalent Refractive Error in Fellow Eye at Enrollment [Number; unit: participants]
  +1.50 to <+2.00 D | 5 | 5 | 10
  +2.00 to <+3.00 D | 6 | 2 | 8
  +3.00 to <+4.00 D | 7 | 9 | 16
  +4.00 D or more | 22 | 17 | 39
Spherical Equivalent Refractive Error in Fellow Eye at Enrollment [Mean (Standard Deviation); unit: diopters] | 3.95 (1.60) | 4.55 (2.28) | 4.22 (1.95)

OUTCOME MEASURES:

1. Primary Outcome: Distribution of 10-week Amblyopic-Eye Visual Acuity
Description: The masked 10-week amblyopic eye visual acuity scores were tabulated for both treatment groups, and included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The primary outcome analysis followed the intent-to-treat principle and included data from 10-week visual acuity exams completed between 8 and 15 weeks (inclusive) with no imputation for missing data.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants
  20/200 | 0 | 1
  20/160 | 2 | 0
  20/125 | 1 | 2
  20/100 | 4 | 0
  20/80 | 5 | 4
  20/63 | 3 | 4
  20/50 | 6 | 6
  20/40 | 11 | 4
  20/32 | 3 | 6
  20/25 | 3 | 5
  20/20 | 1 | 1
  20/16 | 0 | 0

2. Secondary Outcome: Treatment Group Comparison of the Proportion of Participants Who Achieved 20/25 or Better Visual Acuity at 10 Weeks Since Randomization
Description: The proportion of participants who achieved 20/25 or better visual acuity since randomization was computed at the 10-week outcome.
  The secondary outcome analysis was a treatment group comparison of the proportion of participants whose 10-week masked amblyopic eye visual acuity was 20/25 or better since randomization. The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis includes data from participants who completed a 10-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants | 4 | 6

3. Secondary Outcome: Treatment Group Comparison of the Proportion of Participants Who Have Improved by 2 or More logMAR Visual Acuity Lines at 10 Weeks Since Randomization
Description: The proportion of participants who improved at least 2 logMAR lines since randomization was computed at the 10-week outcome.
  The secondary outcome analysis was a treatment group comparison of the proportion of participants whose 10-week masked amblyopic eye visual acuity improved at least 2 logMAR lines since randomization using logistic regression, adjusting for visual acuity at randomization. The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants | 8 | 9
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; Test type: Superiority or Other; p = 0.33, Binomial regression; adjusted for visual acuity at randomization; Risk Difference (RD) = 1, 95% CI 2-sided [-10 to 30]

4. Secondary Outcome: Spectacle Compliance at 10 Weeks by Treatment Group
Description: The distribution of compliance with prescribed treatment was tabulated for the 10-week outcome. Compliance was evaluated as excellent (>75%), good (51%-75%), fair (26%-50%), or poor (<26%) based on discussions with the parent and by reviewing study calendars maintained by the parent, who recorded the frequency of atropine administration.
Time Frame: 10 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  Excellent | 39 | 30
  Good | 1 | 1
  Fair | 0 | 1
  Poor | 0 | 1

5. Secondary Outcome: Average Spectacle Compliance by Treatment Group
Description: The distribution of compliance with prescribed treatment was tabulated for the 10-week outcome and as averaged scores across all study follow-up visits. Compliance was evaluated as excellent (>75%), good (51%-75%), fair (26%-50%), or poor (<26%) based on discussions with the parent and by reviewing study calendars maintained by the parent, who recorded the frequency of atropine administration.
Time Frame: 10 weeks after randomization or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  Excellent | 39 | 30
  Good | 1 | 2
  Fair | 0 | 0
  Poor | 0 | 1

6. Secondary Outcome: Atropine Compliance at 10 Weeks by Treatment Group
Description: as for outcome 4
Time Frame: 10 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  Excellent | 38 | 31
  Good | 2 | 2
  Fair | 0 | 0
  Poor | 0 | 0

7. Secondary Outcome: Average Atropine Compliance by Treatment Group
Description: as for outcome 5
Time Frame: 10 weeks after randomization or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  Excellent | 39 | 29
  Good | 1 | 4
  Fair | 0 | 0
  Poor | 0 | 0

8. Primary Outcome: Mean 10-week Amblyopic-Eye Visual Acuity
Description: The primary outcome analysis was a treatment group comparison of the masked 10-week amblyopic eye visual acuity using an analysis of covariance (ANCOVA) model, adjusting for visual acuity at randomization. The analysis included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
logMAR | 0.42 (0.22) | 0.37 (0.23)
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; The primary analysis was a treatment group comparison of the masked 10-week amblyopic eye visual acuity using an analysis of covariance (ANCOVA) model, adjusting for visual acuity at randomization. The analysis was a 2-sided test for efficacy to test the null hypothesis of no treatment difference, assuming 90% power and a type I error rate of 5%; Test type: Superiority or Other; p = 0.12, ANCOVA; The ANCOVA model included amblyopic eye visual acuity at randomization as an adjustment covariate; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.01 to 0.12] — Positive values favor the Intensified Treatment group

9. Primary Outcome: Distribution of the Change in Amblyopic-Eye Visual Acuity
Description: The change in 10-week amblyopic eye visual acuity scores since randomization was tabulated for both treatment groups, and included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: Randomization to 10 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants
  3 or more lines worse | 0 | 0
  2 lines worse | 1 | 2
  1 line worse | 4 | 3
  No change | 14 | 6
  1 line improved | 12 | 13
  2 lines improved | 7 | 2
  3 or more lines improved | 1 | 7

10. Primary Outcome: Mean Change in Amblyopic-Eye Visual Acuity at 10 Weeks From Randomization
Description: The change in 10-week amblyopic eye visual acuity was computed for both treatment groups and included data from 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) with no imputation for missing data.
  The primary outcome analysis followed the "intent-to-treat" principle. Therefore, data from randomized participants were included in the analysis regardless of whether the assigned treatment was actually received or whether they deviated from treatment against protocol. In addition, randomized participants who were found to be ineligible upon subsequent review of enrollment data were included in the primary outcome analysis.
Time Frame: Randomization to 10 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
logMAR lines | 0.6 (1.1) | 1.1 (1.8)

11. Secondary Outcome: Distribution of Interocular Difference at 12-week Exam
Description: Distribution of Interocular Difference Between Eyes at 12-week Exam
Time Frame: 12 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants
  0 or less lines | 3 | 2
  1 line | 2 | 2
  2 lines | 6 | 8
  3 lines | 6 | 8
  4 lines | 5 | 4
  5 lines | 5 | 5
  6 or more lines | 12 | 4

12. Secondary Outcome: Mean Interocular Difference at 12-week Exam
Description: Mean Interocular Difference Between Eyes at 12-week Exam
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
logMAR lines | 4.3 (2.6) | 3.3 (2.0)

13. Secondary Outcome: Distribution of 12-week Fellow-Eye Visual Acuity
Description: Following the 10-week primary outcome exam, participants discontinued the randomized treatment and returned 2 weeks later for a 12-week visit to measure off-treatment fellow-eye visual acuity.
Time Frame: 12 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  20/40 | 1 | 0
  20/32 | 0 | 4
  20/25 | 10 | 7
  20/20 | 19 | 14
  20/16 | 10 | 8

14. Secondary Outcome: Mean Fellow-Eye Visual Acuity at 12-week Exam
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
logMAR | 0.01 (0.09) | 0.02 (0.10)

15. Secondary Outcome: Distribution of Change in Fellow-Eye Visual Acuity at 12 Weeks From Randomization
Time Frame: 12 weeks after randomization
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  3 or more lines worse | 1 | 0
  2 lines worse | 0 | 0
  1 line worse | 1 | 2
  No change | 23 | 22
  1 line improved | 12 | 7
  2 lines improved | 3 | 2
  3 or more lines improved | 0 | 0

16. Secondary Outcome: Mean Change in Fellow-Eye Visual Acuity at 12 Weeks From Randomization
Time Frame: 12 weeks after randomization
Measure: Mean (Standard Deviation); unit: change in lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
change in lines | 0.4 (0.9) | 0.3 (0.7)
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; A treatment group difference in fellow-eye visual acuity change at the 12-week exam was evaluated using an ANCOVA model, adjusting for the fellow-eye visual acuity at randomization; Test type: Superiority or Other; p = 0.55, ANCOVA; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.23 to 0.43]

17. Secondary Outcome: Distribution of Baseline Characteristics at the 10-week Outcome
Description: The number of participants was tabulated by treatment group within categorical levels of prespecified baseline subgroup factors for participants with 10-week visual acuity exams completed between 8 to 15 weeks (inclusive) according to principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis included participants who completed 10-week exams between 8 and 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants
  Gender: Female | 21 | 19
  Gender: Male | 18 | 14
  Race/Ethnicity: White (non-Hispanic) | 32 | 29
  Race/Ethnicity: Non-White/Hispanic | 7 | 4
  Age at randomization: 3 to <4 years | 5 | 4
  Age at randomization: 4 to <5 years | 7 | 6
  Age at randomization: 5 to <6 years | 9 | 9
  Age at randomization: 6 to <7 years | 7 | 5
  Age at randomization: 7 years or older | 11 | 9
  Amblyopic-eye VA at randomization: 20/80 or worse | 11 | 10
  Amblyopic-eye VA at randomization: 20/63 | 9 | 8
  Amblyopic-eye VA at randomization: 20/50 | 7 | 8
  Amblyopic-eye VA at randomization: 20/40 or better | 12 | 7
  Cause of amblyopia: Strabismus | 8 | 13
  Cause of amblyopia: Anisometropia | 10 | 6
  Cause of amblyopia: Combined mechanism | 21 | 14
  Atropine duration prior to randomization:12-<15wks | 11 | 5
  Atropine duration prior to randomization:15-<21wks | 6 | 9
  Atropine duration prior to randomization:21-<27wks | 12 | 9
  Atropine duration prior to randomization:27-84 wks | 10 | 10
  Fellow-eye SE RE at enrollment: <+3.00 Diopters(D) | 10 | 7
  Fellow-eye SE RE at enrollment: +3.00 to <+4.50 D | 12 | 13
  Fellow-eye SE RE at enrollment: +4.50 to +6.00 D | 12 | 4
  Fellow-eye SE RE at enrollment: >+6.00 D | 5 | 9

18. Secondary Outcome: Mean Amblyopic Eye Visual at Randomization According to Baseline Characteristics for 10-week Outcome
Description: Mean amblyopic eye visual acuity at randomization was computed by treatment group within categorical levels of prespecified baseline subgroup factors. The analysis included data from participants with 10-week exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: The analysis included participants who completed 10-week exams between 8 and 15 weeks (inclusive) according to the principles of the primary outcome analysis.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
logMAR
  Gender: Female | 0.51 (0.19) | 0.46 (0.14)
  Gender: Male | 0.45 (0.19) | 0.51 (0.19)
  Race/Ethnicity: White (non-Hispanic) | 0.50 (0.19) | 0.49 (0.17)
  Race/Ethnicity: Non-White/Hispanic | 0.41 (0.18) | 0.43 (0.05)
  Age at randomization: 3 to <4 years | 0.58 (0.22) | 0.48 (0.17)
  Age at randomization: 4 to <5 years | 0.50 (0.13) | 0.58 (0.23)
  Age at randomization: 5 to <6 years | 0.46 (0.21) | 0.42 (0.10)
  Age at randomization: 6 to <7 years | 0.43 (0.18) | 0.50 (0.12)
  Age at randomization: 7 years or older | 0.48 (0.21) | 0.48 (0.18)
  Cause of amblyopia: Strabismus | 0.48 (0.23) | 0.46 (0.16)
  Cause of amblyopia: Anisometropia | 0.42 (0.13) | 0.35 (0.11)
  Cause of amblyopia: Combined mechanism | 0.51 (0.20) | 0.56 (0.15)
  Atropine duration prior to randomization:12-<15wks | 0.54 (0.23) | 0.38 (0.11)
  Atropine duration prior to randomization:15-<21wks | 0.53 (0.23) | 0.51 (0.18)
  Atropine duration prior to randomization:21-<27wks | 0.43 (0.12) | 0.53 (0.12)
  Atropine duration prior to randomization:27-84 wks | 0.46 (0.18) | 0.47 (0.19)
  Fellow-eye SE RE at enrollment: <+3.00 Diopters(D) | 0.41 (0.20) | 0.49 (0.20)
  Fellow-eye SE RE at enrollment: +3.00 to <+4.50 D | 0.50 (0.18) | 0.51 (0.16)
  Fellow-eye SE RE at enrollment: +4.50 to +6.00 D | 0.53 (0.17) | 0.45 (0.24)
  Fellow-eye SE RE at enrollment: >+6.00 D | 0.48 (0.25) | 0.47 (0.11)

19. Secondary Outcome: Treatment Comparison of Mean Amblyopic Eye Visual Acuity Change at 10-weeks According to Baseline Characteristics
Description: A treatment comparison of mean amblyopic eye visual acuity change since randomization was performed at the 10-week outcome according to categorical levels of prespecified baseline subgroup factors. The analysis included data from participants with 10-week exams completed between 8 to 15 weeks (inclusive) according to the principles specified in the primary outcome analysis.
Time Frame: 10 weeks after randomization
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
logMAR lines
  Gender: Female | 0.2 (1.0) | 1.2 (1.6)
  Gender: Male | 1.0 (1.0) | 1.1 (2.0)
  Race/Ethnicity: White (non-Hispanic) | 0.5 (1.1) | 1.1 (1.8)
  Race/Ethnicity: Non-White/Hispanic | 0.9 (1.2) | 1.0 (2.2)
  Age at randomization: 3 to <4 years | 0.2 (0.8) | 1.3 (1.3)
  Age at randomization: 4 to <5 years | 04 (1.5) | 0.7 (2.4)
  Age at randomization: 5 to <6 years | 0.8 (1.3) | 1.2 (1.4)
  Age at randomization: 6 to <7 years | 0.3 (0.5) | 2.4 (2.0)
  Age at randomization: 7 years or older | 0.9 (0.9) | 0.6 (1.7)
  Amblyopic-eye VA at randomization: 20/80 or worse | 0.5 (0.7) | 1.0 (2.4)
  Amblyopic-eye VA at randomization: 20/63 | 0.4 (1.3) | 1.5 (1.7)
  Amblyopic-eye VA at randomization: 20/50 | 1.0 (1.3) | 1.3 (1.7)
  Amblyopic-eye VA at randomization: 20/40 or better | 0.5 (1.1) | 0.7 (1.0)
  Cause of amblyopia: Strabismus | 0.1 (1.1) | 1.7 (1.8)
  Cause of amblyopia: Anisometropia | 0.8 (0.9) | 1.0 (1.9)
  Cause of amblyopia: Combined mechanism | 0.7 (1.1) | 0.6 (1.6)
  Atropine duration prior to randomization:12-<15wks | 1.1 (0.7) | 1.2 (1.8)
  Atropine duration prior to randomization:15-<21wks | -0.3 (1.0) | 1.7 (2.2)
  Atropine duration prior to randomization:21-<27wks | 0.6 (1.3) | 1.2 (1.5)
  Atropine duration prior to randomization:27-84 wks | 0.6 (0.8) | 0.5 (1.6)
  Fellow-eye SE RE at enrollment: <+3.00 Diopters(D) | 0.7 (1.3) | 1.0 (2.7)
  Fellow-eye SE RE at enrollment: +3.00 to <+4.50 D | 0.7 (1.2) | 1.0 (1.2)
  Fellow-eye SE RE at enrollment: +4.50 to +6.00 D | 0.4 (0.9) | 1.3 (2.6)
  Fellow-eye SE RE at enrollment: >+6.00 D | 0.6 (1.1) | 1.3 (1.4)

20. Secondary Outcome: Distribution of Amblyopic-Eye Visual Acuity at Best Outcome Visit
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The distribution of best post-randomization (10 weeks or later) visual acuity scores in the amblyopic eye was tabulated for both treatment groups using the initial visual acuity score (if a retest was obtained.)
Time Frame: 10 weeks after randomization or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  20/200 | 0 | 1
  20/160 | 2 | 0
  20/125 | 1 | 0
  20/100 | 3 | 1
  20/80 | 6 | 1
  20/63 | 1 | 4
  20/50 | 8 | 5
  20/40 | 10 | 3
  20/32 | 3 | 10
  20/25 | 5 | 5
  20/20 | 1 | 3
  20/16 | 0 | 0

21. Secondary Outcome: Mean Amblyopic-Eye Visual Acuity at Best Outcome Visit
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. A treatment comparison of mean amblyopic eye visual acuity at the visit of best post-randomization visual acuity (10 weeks or later) was performed using an analysis of covariance, adjusting for amblyopic eye visual acuity at randomization.
Time Frame: 10 weeks after randomization or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
logMAR | 0.40 (0.23) | 0.29 (0.22)

22. Secondary Outcome: Distribution of Change in Amblyopic-Eye Visual Acuity From Randomization to Best Outcome Visit
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The distribution of change in best post-randomization (10 weeks or later) visual acuity in the amblyopic eye since randomization was tabulated for both treatment groups using the initial visual acuity score (if a retest was obtained.)
Time Frame: Randomization to 10 weeks or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  3 or more lines worse | 0 | 0
  2 lines worse | 1 | 1
  1 line worse | 4 | 3
  No change | 12 | 3
  1 line improved | 12 | 6
  2 lines improved | 9 | 6
  3 or more lines improved | 2 | 14

23. Secondary Outcome: Mean Change in Amblyopic-Eye Visual Acuity at Best Outcome Visit
Description: Participants in both groups who have improved by one or more lines from randomization to the 10-week outcome exam will continue in the study and visits will occur every 10 weeks until no improvement of one or more lines from the previous visit. The mean change in amblyopic eye visual acuity since randomization was computed for both treatment groups based on the visit of best post-randomization visual acuity (10 weeks or later) using the initial visual acuity score (if a retest was obtained.)
Time Frame: 10 weeks after randomization or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Population: The analysis includes data from participants who completed the 10-week exam and/or a later visit.
Measure: Mean (Standard Deviation); unit: logMAR lines
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 30
logMAR lines | 0.8 (1.2) | 1.9 (1.8)

24. Secondary Outcome: Treatment Group Comparison of the Proportion of Participants Who Have Improved by 2 or More logMAR Visual Acuity Lines Based on Visual Acuity at Best Outcome Visit
Time Frame: 10 weeks after randomization or later (until no further VA improvement, up to maximum of 84 weeks for one subject)
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 39 | 33
participants | 11 | 20

25. Secondary Outcome: Distribution of Randot Preschool Stereoacuity Score at 12 Weeks
Description: Distribution of Randot Preschool Stereoacuity Score at 12 Weeks; Participants with a Randot Preschool test of >800 seconds of arc were classified as having a stereoacuity of 3000 seconds of arc if the Titmus fly test was positive or as nil if the Titmus fly test was negative.
Time Frame: 12 weeks after randomization
Population: The analysis includes all participants who completed the 12-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 40 | 33
participants
  Failed pretest | 4 | 2
  >800 arcsec: Nil | 7 | 10
  >800 arcsec: 3000 arcsec | 14 | 12
  800 arcsec | 7 | 3
  400 arcsec | 4 | 3
  200 arcsec | 0 | 1
  100 arcsec | 1 | 1
  60 arcsec | 2 | 1
  40 arcsec | 1 | 0
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; The distribution of 12-week Randot Preschool Stereoacuity scores was compared between treatment groups using a Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.23, Wilcoxon (Mann-Whitney)

26. Secondary Outcome: Distribution of Randot Preschool Stereoacuity Scores at 12 Weeks for Participants With Anisometropic Amblyopia
Time Frame: 12 weeks after randomization
Population: The analysis includes participants with anisometropic amblyopia (no strabismus) who completed the 12-week exam.
Measure: Number; unit: participants
Arm/Group | Control | Intensified Treatment
Number analyzed (Participants) | 10 | 6
participants
  Failed pretest | 0 | 0
  >800 arcsec: Nil | 1 | 1
  >800 arcsec: 3000 arcsec | 2 | 2
  800 arcsec | 3 | 1
  400 arcsec | 2 | 0
  200 arcsec | 0 | 0
  100 arcsec | 0 | 1
  60 arcsec | 1 | 1
  40 arcsec | 1 | 0
Statistical Analysis 1: Comparison: Control vs Intensified Treatment; [analysis description as in outcome 25, analysis 1]; Test type: Superiority or Other; p = 0.66, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Control | Intensified Treatment
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/33
Other Adverse Events (participants affected / at risk) | 5/40 | 9/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control (N=40) | Intensified Treatment (N=33)
Light Sensitivity (Eye disorders) | 1 | 6
New ocular deviation or worsening of preexisting deviation by at least 10 PD (Eye disorders) | 4 | 3

LIMITATIONS AND CAVEATS:
A potential study limitation is that compliance with patching was based on discussions with the parent and by reviewing study calendars maintained by the parent, which not an objective measure of compliance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No